CLINICAL TRIAL: NCT04455906
Title: Mechanisms of Increased Disease Severity in AD Patients With the IL-4Ra R576 Polymorphism
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Wanda Phipatanakul, Professor of Pediatrics, Director Asthma Research Center, Harvard Medical School (HMS and HSDM)
Other Study IDs: IRB-P00035467
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, skin tape, biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This protocol is primarily looking to see if the IL-4Ra R576 polymorphism is associated with increased clinical, immunological and microbial markers of disease activity in patients with Atopic dermatitis.

DETAILED DESCRIPTION:
For this study, participants ages 6-65 years, who have atopic dermatitis and don't have any of the exclusion criteria will be invited to participate in the study. There will be a 1 time visit where questionnaires, blood draw, skin swab and skin biopsies will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥6 to 65 yrs of age
2. Meet AD Standard Diagnostic Criteria

Exclusion Criteria:

1. Enrollment in another clinical trial
2. Hypersensitivity to an agent used for the skin decolonization protocol
3. Use within 4 weeks of systemic treatment with immunosuppressive/immunomodulating drugs (corticosteroids, cyclosporine, mycophenolate, JAK inhibitors, azathioprine, methotrexate)
4. Phototherapy for AD within 4 weeks
5. Treatment with biologics (dupilumab, omalizumab, benralizumab, etc) within sixteen weeks
6. Use of topical steroids, topical calcineurin inhibitors or crisaborale within 7 days
7. Bleach baths within 7 days of the first Visit
8. Use of oral or topical antibiotics within 21 days of the beginning of the study
9. Asthmatics receiving more than 500 μg per day of inhaled corticosteroids
10. History of (HIV, hepatitis B, hepatitis C, tuberculosis malignancy
11. Skin comorbidities that may interfere with assessments: psoriasis, cutaneous T Cell lymphoma,,
12. Severe ongoing medical illnesses e.g. cardiovascular, renal disease, autoimmune disease.
13. Febrile illness at time of visits
14. Suspected immune deficiency or family history of primary immunodeficiency

Ages: 6 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: atopic dermatitis
Sampling Method: Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
atopic dermatitis severity | baseline, only 1 time point
  validated assessment EASI score

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Phipatanakul, MD. MS., Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States